CLINICAL TRIAL: NCT02768012
Title: Mindfulness for Antidepressant-induced Sexual Symptoms
Acronym: MASS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Potential participants to date all had etiological factors for their sexual dysfunction additional to the antidepressant. Thus they all had exclusion criterior
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rosemary Basson, Clinical Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H15-02707
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Other Substance Induced Sexual Dysfunction
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mindfulness-based cognitive therapy (Active Comparator): The practice of mindfulness will be followed plus the basics of cognitive therapy given in small group format.
  Interventions: Behavioral: mindfulness-based cognitive therapy
- waitlist (No Intervention): Women diagnosed with AISD randomised to wait list will receive no active treatment during the trial period.

INTERVENTIONS:
Behavioral: mindfulness-based cognitive therapy — Six two-hour small group sessions (6-9 participants) will be administered over 8 weeks focusing on MBCT. The intervention follows a written protocol to ensure fidelity of delivery. Participants will receive detailed manuals summarizing session content and home assignments (HAs), including mindfulness practices, audio versions of which will be available on an internet link.
  Arms: mindfulness-based cognitive therapy

SUMMARY:
Antidepressant-induced sexual dysfunction (AISD) affects the majority of women taking antidepressants and reduces medication compliance: however there is a paucity of evidence-based strategies for the management of this condition. Mindfulness-based cognitive therapy (MBCT) has been shown to be effective in the treatment of non-antidepressant-induced sexual dysfunction and may be beneficial in the treatment of AISD. The investigators propose a randomized, controlled, proof-of-principle trial to establish preliminary evidence of efficacy of MBCT in AISD and to inform the design of a larger trial to evaluate its effectiveness

DETAILED DESCRIPTION:
The investigators propose a randomized, controlled, proof-of-principle trial to establish preliminary evidence of efficacy of MBCT in AISD and to inform the design of a larger trial to evaluate its effectiveness.

2. Objectives

1. To provide preliminary evidence of efficacy of MBCT in the management of AISD.
2. To establish the feasibility of conducting a larger RCT of MBCT in AISD by assessing recruitment, attendance and retention rates.
3. To determine the minimal clinically important difference (MCID) for the Changes in Sexual Functioning Questionnaire (CSFQ-14) and the Female Sexual Function Index (FSFI).
4. To gain initial estimates of variability for sample size calculation for future trials of interventions in this patient population.

Study design: Randomized, controlled, parallel-group trial. There will be two treatments: a mindfulness-based group intervention and a wait-list control. Randomization will be 2:1 (MBCT: WLC). This will be an open-label single center study.

Procedures: Ethics approval will be obtained from the University of British Columbia (UBC) Clinical Research Ethics Board (CREB). Upon referral to the UBC sexual medicine clinic, women are assessed by a clinician with expertise in sexual medicine. Those diagnosed with AISD, and deemed as likely eligible, are informed about the study and invited to meet with the study coordinator who will assess study criteria and provide more detail about the study procedures. If the patient agrees to participation, she will first read the consent form and accept it. The coordinator will then email her a direct link to the online survey. Upon accessing the link, she will then be routed to the online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* participants need to be:

  1. referred to the Sexual Medicine Clinic
  2. women 19 years of age or older
  3. fulfilling the DSM-5 criteria for clinical diagnosis of AISD for at least 4 weeks, confirmed by Changes in Sexual Functioning Questionnaire (CSFQ-14) total score of 41 or below
  4. on a therapeutic dose of antidepressant for at least 8 weeks and on a stable dose for at least 4 weeks
  5. in clinical remission from depression and/or anxiety, confirmed by a Patient Health Questionnaire (PHQ-9) score of less than 5, and a Generalized Anxiety Disorder-7 (GAD-7) score of less than 10, respectively
  6. willing to commit to adhere to their antidepressant regimen for the duration of the trial (20 weeks) unless medically contraindicated
  7. willing to commit to attend to all group sessions, homework assignments, and questionnaires
  8. the referring physician commits to continued provision of mental health care throughout the study

Exclusion Criteria:

1. history of SD prior to being started on current antidepressant except SD secondary to clinical depression, or AISD
2. chronic pain with intercourse not relieved with lubricants
3. primary psychiatric disorder other than a depressive or anxiety disorder
4. alcohol/substance abuse
5. general medical illnesses known to impair sexual function including but not limited to cancer, neurological, endocrine, renal, and cardiovascular conditions
6. non-antidepressant medication induced SD (70)
7. receiving other concurrent pharmacological or psychological interventions for SD
8. positive screen for borderline personality disorder, due to the high prevalence of sexual difficulties (70, 71), and the potential destabilizing effect of mindfulness meditation in those affected (72)
9. previous formal practice of mindfulness meditation.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
group difference on change in CSFQ-14 score after intervention | 18 months
  The researchers will calculate an 80% confidence interval for the between group difference on change in CSFQ-14 score pre to post intervention using a linear mixed model that includes treatment, time and time-by-treatment as fixed effects and patient as a random effect. If the confidence interval excludes 0 the researchers will consider this preliminary evidence of efficacy.

SECONDARY OUTCOMES:
Estimation of the minimal clinically important improvement | 18 months
  At treatment completion (8 weeks) patients will be asked to assess their response to MBCT treatment on a five-point descriptive scale (none = no good at all, treatment was ineffective; poor = some effect but unsatisfactory; fair = reasonable effect but could be better; good = satisfactory effect but still some problems; excellent = ideal response, sexual dysfunction gone). The minimal clinically important improvement for the CSFQ-14 and the FSFI will be determined from the group reporting a "good" response following established methods.

IPD SHARING:
Plan to Share IPD: No